CLINICAL TRIAL: NCT04021810
Title: Combination Therapy Associating CPAP and Mandibular Advancement Device ( MAD) in Obstructive Sleep Apnea (OSA) Low CPAP Compliers: A Randomized Controlled Trial
Brief Title: Combination Therapy Associating CPAP and Mandibular Advancement Device in OSA
Acronym: PPC-OAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of faisability
Sponsor: University Hospital, Grenoble (Other)
Collaborators: ONIRIS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.350
Record Dates: First submitted 2019-06-18; First posted 2019-07-16 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea Syndrome; Hypertension
Keywords: Sleep Apnea; CPAP; Mandibular Advancement Device; Arterial Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure; Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPAP only (Active Comparator): Obstructive sleep apnea patients with CPAP treatment only
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) and patient education
- Mandibular Advancement Device only (Active Comparator): Obstructive sleep apnea patients with Mandibular Advancement Device only
  Interventions: Device: Mandibular Advancement Device
- CPAP + Mandibular Advancement Device (Experimental): Obstructive sleep apnea patients with combined CPAP and Mandibular Advancement Device
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) and patient education; Device: Mandibular Advancement Device

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) and patient education — Mask connected to a pump (CPAP machine) that forces air into the nasal passages at pressures high enough to overcome obstructions in the airways. Plus patient education.
  Arms: CPAP + Mandibular Advancement Device; CPAP only
Device: Mandibular Advancement Device — Adjustable oral prosthesis which retains the lower mandible in an anterior position, thus limiting sleep apneas
  Arms: CPAP + Mandibular Advancement Device; Mandibular Advancement Device only

SUMMARY:
The aim of this study is to evaluate the efficacy of a combination of Continuous Positive Airway Pressure (CPAP) and a Mandibular Advancement Device (MAD) on nocturnal Blood Pressure control in hypertensive patients in obstructive sleep apnea low CPAP compliers (less than 4 hours per night).

Hypertensive patients demonstrating low CPAP adherence will be selected during a screening visit; they will be then randomized to one of the three following arms: Education to CPAP ("CPAP only"), Treatment by a MAD ("MAD only") or a combination of both CPAP and MAD ("CPAP+MAD"). Mean systolic, diastolic, diurnal and nocturnal blood pressure will be assessed during 24-h Ambulatory Blood Pressure monitoring, before and after a 3-month treatment intervention. Biological laboratory parameters, patients reported outcomes (daytime sleepiness and Quality of Life), will also be evaluated before and after 3 months of treatment.

DETAILED DESCRIPTION:
The aim of this study is to test the efficacy of a combination of Continuous Positive Airway Pressure (CPAP) treatment and a Mandibular Advancement Device (MAD) on the control of nocturnal Blood Pressure over a 3-month period in hypertensive obstructive sleep apnea being low CPAP compliers.

This is a prospective, randomized, open-label and multi-centric study. The investigators plan to include 105 hypertensive patients demonstrating low CPAP adherence (less than 4 hours per night). Patients will be randomly assigned to one of the following treatments: Education for improving CPAP adherence ('CPAP Only' group: patients will continue their CPAP treatment and be supported by regular coaching aimed at increasing their compliance to treatment); Mandibular Advancement Device ('MAD Only' group: patients will switch their treatment from CPAP to a MAD); a combination of CPAP and MAD ('CPAP + MAD' group: patients will be treated by both devices used simultaneously).

The duration of the study is 3 months. At the selection visit, patients will undergo a polysomnography/respiratory polygraphy followed by 24h- Ambulatory Blood Pressure Monitoring, PROMs (Quality of Life, Epworth Sleepiness Score) and a blood sample for biological parameters analysis. Patients will be then randomized to one of the three groups. Patients assigned to the 'CPAP only group' will be contacted by the homecare provider to arrange coaching sessions in order to improve their compliance to CPAP (phone calls and/or home visits). Patients assigned to the 'MAD Only group' will be proposed a Mandibular Advancement Device. Patients assigned to the 'CPAP+MAD group' will have both CPAP (with coaching) and a MAD.

After a 3-month treatment period, the same measurements (24h-Ambulatory Blood pressure, polysomnography/respiratory polygraphy, questionnaires, and blood sample analysis) will be repeated to compare efficacy of the 3 interventions. Tolerance (number of adverse events) and adherence to treatments will also be assessed.

The 'CPAP+MAD' group will be compared to the other two groups in order to evaluate the benefit of the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Arterial Hypertension (Clinical Blood Pressure > 140/90 mmHg or patient under medication with nocturnal hypertension seen in the Ambulatory Blood Pressure Measurement)
* Severe obstructive sleep apnea syndrome, treated by CPAP for more than 6 months and less than 5 years, with a compliance <4h/night
* No contraindication to a treatment by Mandibular Advancement Device
* Ability to understand study procedures and signed informed consent
* Covered by French social security system or equivalent

Exclusion Criteria:

* Central Obstructive Apnea (>20% Central Apneas/Hypopneas)
* Pregnant or breastfeeding womens
* Prisoners or persons who require protection by the law
* Persons within the exclusion period of another study
* Contraindication to a mandibular advancement device (oral-dental pathology, pathology of the temporo-mandibular articulation, poor periodontal status)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Nightime Mean Blood Pressure | 3 months
  Difference in nighttime Mean Blood Pressure before and after treatment, measured by ambulatory blood pressure

SECONDARY OUTCOMES:
Other 24h ambulatory blood pressure measurements | 3 months
  24h ambulatory blood pressure measurements (systolic, diastolic and mean, diurnal and nocturnal) before and after treatment
Blood Pressure Variability | 3 months
  Blood Pressure variability before and after treatment, measured by ambulatory blood pressure measurements
Percent Dippers/dipping phenotypes | 3 months
  Percentage of dipper patients (>10% drop in nocturnal Blood Pressure compared with daytime BP)
3-days home Blood Pressure measurements (systolic, diastolic) | 3 months
  self-measurement of Systolic and Diastolic Blood Pressure, measured over 3 days, twice a day, before and after interventions
Epworth Score | 3 months
  Score on the Epworth Sleepiness Questionnaire, before and after treatment. The ESS is a self-administered questionnaire with 8 questions. Patients are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 sub-item scores( 0-3) can range from 0 to 24. The higher the ESS score the greater the likelihood that the person has daytime sleepiness.
Quality of Life score | 3 months
  Score on the Quality Of Life Questionnaire SF12, before and after treatment. The SF-12 is a self-administered short survey with 12 questions assessing quality of life. The questions are combined, scored, and weighted to create two subscales (mental and social score and physical score) that provide glimpses into health-related quality of life. The lower the scores the more disability.
Serum concentration of Cholesterol | 3 months
  Serum concentration of low-density lipoprotein cholesterol (LPL-C) and high-density lipoprotein cholesterol (HDL-C), before and after treatment.
Serum concentration of Triglycerides | 3 months
  Serum concentration of Triglyceride, before and after treatment
Concentration of fasting Glucose | 3 months
  Concentration of fasting glucose, before and after treatment
Amount of HbA1C | 3 months
  Amount of HbA1c, before and after treatment
Incidence of adverse events related to the treatment | 3 months
  Number of adverse events related to the treatment during the 3-month period
Compliance to treatment(s) | 3 months
  Use of the device(s) defined by number of hour per night and number of night per week
Efficacy determined by comparison of Apnea-Hypopnea Index (AHI), number of central and obstructive apneas and hypopneas, before and after treatment | 3 months
  AHI, central and obstructive apneas and hyponeas index, measured by polysomnography or polygraphy, before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, Pr, PhD, Principal Investigator — University Hospital, Grenoble
Locations (4):
- France (4):
  - Nouvelle Clinique Bel Air, Bordeaux
  - University Hospital Grenoble, Grenoble
  - University Hospital Montpellier, Montpellier
  - Cabinet Médical, Perpignan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Result] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Result] Kendzerska T, Gershon AS, Hawker G, Leung RS, Tomlinson G. Obstructive sleep apnea and risk of cardiovascular events and all-cause mortality: a decade-long historical cohort study. PLoS Med. 2014 Feb 4;11(2):e1001599. doi: 10.1371/journal.pmed.1001599. eCollection 2014 Feb. PMID 24503600
- [Result] Bailly S, Destors M, Grillet Y, Richard P, Stach B, Vivodtzev I, Timsit JF, Levy P, Tamisier R, Pepin JL; scientific council and investigators of the French national sleep apnea registry (OSFP). Obstructive Sleep Apnea: A Cluster Analysis at Time of Diagnosis. PLoS One. 2016 Jun 17;11(6):e0157318. doi: 10.1371/journal.pone.0157318. eCollection 2016. PMID 27314230
- [Result] Levy P, Kohler M, McNicholas WT, Barbe F, McEvoy RD, Somers VK, Lavie L, Pepin JL. Obstructive sleep apnoea syndrome. Nat Rev Dis Primers. 2015 Jun 25;1:15015. doi: 10.1038/nrdp.2015.15. PMID 27188535
- [Result] Bratton DJ, Gaisl T, Schlatzer C, Kohler M. Comparison of the effects of continuous positive airway pressure and mandibular advancement devices on sleepiness in patients with obstructive sleep apnoea: a network meta-analysis. Lancet Respir Med. 2015 Nov;3(11):869-78. doi: 10.1016/S2213-2600(15)00416-6. Epub 2015 Oct 20. PMID 26497082
- [Result] Pepin JL, Tamisier R, Baguet JP, Lepaulle B, Arbib F, Arnol N, Timsit JF, Levy P. Fixed-pressure CPAP versus auto-adjusting CPAP: comparison of efficacy on blood pressure in obstructive sleep apnoea, a randomised clinical trial. Thorax. 2016 Aug;71(8):726-33. doi: 10.1136/thoraxjnl-2015-207700. Epub 2016 Apr 18. PMID 27091542
- [Result] Pepin JL, Tamisier R, Barone-Rochette G, Launois SH, Levy P, Baguet JP. Comparison of continuous positive airway pressure and valsartan in hypertensive patients with sleep apnea. Am J Respir Crit Care Med. 2010 Oct 1;182(7):954-60. doi: 10.1164/rccm.200912-1803OC. Epub 2010 Jun 3. PMID 20522795
- [Result] Malhotra A, Orr JE, Owens RL. On the cutting edge of obstructive sleep apnoea: where next? Lancet Respir Med. 2015 May;3(5):397-403. doi: 10.1016/S2213-2600(15)00051-X. Epub 2015 Apr 14. PMID 25887980
- [Result] Bratton DJ, Gaisl T, Wons AM, Kohler M. CPAP vs Mandibular Advancement Devices and Blood Pressure in Patients With Obstructive Sleep Apnea: A Systematic Review and Meta-analysis. JAMA. 2015 Dec 1;314(21):2280-93. doi: 10.1001/jama.2015.16303. PMID 26624827
- [Result] Mokhlesi B, Hagen EW, Finn LA, Hla KM, Carter JR, Peppard PE. Obstructive sleep apnoea during REM sleep and incident non-dipping of nocturnal blood pressure: a longitudinal analysis of the Wisconsin Sleep Cohort. Thorax. 2015 Nov;70(11):1062-9. doi: 10.1136/thoraxjnl-2015-207231. Epub 2015 Aug 25. PMID 26307037